CLINICAL TRIAL: NCT06261450
Title: Effect of CBD on the GABAergic System in Patients with Fragile X Syndrome.
Brief Title: Effect of CBD on the Brain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Jazz Pharmaceuticals (Industry); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Francois Corbin, Full professor, Department of biochemistry, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2020-3424; 236114 (Other: Health Canada); 202010PJT-451514 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-01-26; First posted 2024-02-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Fragile X Syndrome
Keywords: MRI; Cannabidiol; GABA; FXS; MRS; TMS
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a double-blind-crossover placebo control comparing the acute effect of oral CBD in patients with FXS to controls.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization and dispensing of active and control will be conducted by the research center pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBD first (Experimental): A single dose of CBD dose administered followed by a dose of placebo 3 weeks later.
  Interventions: Drug: CBD Oral Solution (eCBD system Target); Drug: Placebo
- Placebo first (Experimental): A single dose of placebo dose administered followed by a dose of CBD 3 weeks later.
  Interventions: Drug: CBD Oral Solution (eCBD system Target); Drug: Placebo

INTERVENTIONS:
Drug: CBD Oral Solution (eCBD system Target) — Participants receive orally 6 ml of CBD Oral Solution (100 mg / ml; 60 mg / kg; max 600 mg of CBD) followed by 6 ml of a placebo composed of the inactive ingredients of CBD Oral Solution 3 weeks later.
Drug: Placebo — Participants receive orally 6 ml of a placebo composed of the inactive ingredients of CBD Oral Solution followed by 6 ml of Oral CBD Solution (100 mg / ml; 60 mg / kg; max 600 mg of CBD)

SUMMARY:
This proposal focuses on the therapeutic relevance of the endocannabinoid (eCB) system for the treatment of Fragile-X syndrome (FXS), the primary hereditary cause of autism spectrum disorder (ASD). Although most individuals with FXS have moderate to severe intellectual disability (ID), caregivers are mainly concerned about aggressive behavior and anxiety problems, hallmark features of the condition. Concurrent lines of evidence suggest that targeting the endocannabinoid (eCB) system by administration of cannabidiol (CBD) could upregulate GABAergic functions and correct inhibitory deficits presumed responsible for the neuropsychiatric phenotype of FXS. However, the eCB system and its effect on the brain remains unexplored in FXS patients. This clinical trial aims to define the therapeutic relevance of the eCB system for FXS using a multimodal neuroimaging approach to finely characterize the acute effects of oral CBD on the principal inhibitory neurotransmitter system (GABA) in a large cohort of FXS patients.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for FXS participants will include:

* age between 7 and 55 years, molecular diagnosis of FXS,
* intelligence quotient (IQ) <70,
* aberrant behavior questionnaire score (ABC-C) > 20,
* <3 psychoactive drugs, drug stable for > 3 months.

Eligibility criteria for the control group:

* 18 and 55 years old,
* be in good general health, with no history of neurological or psychiatric disorders.

Eligibility Criteria for all Participants:

* A minimum weight of 60 kg;
* no history of liver problems (A complete blood profile to measure liver enzyme levels (bilirubin, aspartate aminotransferase (AST), argininosuccinate lyase (ASL), alanine transaminase (ALT), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT)) will be obtained before randomization for all participants).

Exclusion Criteria:

* The presence of an absolute contraindication to the use of TMS and MRI / MRS (ie presence of metal in the head).
* Individuals with ALT / ASL levels greater than 3 times the upper normal baseline, or if bilirubin exceeds 2 times the upper baseline,

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Short Intracortical Inhibition | Comparison between pre and 2 hours post administration of Oral CBD solution and placebo
  Transcranial Magnetic Stimulation (TMS)-derived measure of Intracortical inhibition: The degree of decrease of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 70% of resting motor threshold) 2-4 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 millivolt (mV), approximately 120% of resting motor threshold)

SECONDARY OUTCOMES:
Intracortical Facilitation | Comparison between pre and 2 hours post administration of Oral CBD solution and placebo
  TMS-derived measure of Intracortical Facilitation: The degree of increase of peak-to-peak motor evoked potential (MEP) amplitude induced by the administration of a conditioning stimulus (set at 80% of resting motor threshold) 12-24 ms before the test stimulus (stimulation intensity required to produce an MEP of 1 mV, approximately 120% of resting motor threshold).
Gaba concentration levels | Comparison between pre and 2 hours post administration of Oral CBD solution and placebo
  Estimation of GABA concentrations in the brain from magnetic resonance spectroscopy (MRS)

IPD SHARING:
Plan to Share IPD: No